CLINICAL TRIAL: NCT03051828
Title: Practice of Fencing in Breast Cancer Care
Brief Title: Physical Evaluation and Quality of Life in the Practice of Fencing in Breast Cancer Support
Acronym: ESCRIME
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0115
Record Dates: First submitted 2016-09-13; First posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: fencing, cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fencing and patients with breast cancer: patients operated for breast cancer followed at the Hospital Rene Dubos
  Interventions: Procedure: fencing

INTERVENTIONS:
Procedure: fencing — No intervention: practice fencing

SUMMARY:
The data collection of physical evaluations after regular practice of the fencing at patients having surgically been treated for breast cancer highlighted encouraging results both on the functional drawing, and on the improvement of the quality of life.

DETAILED DESCRIPTION:
Recent scientific works show that a regular physical activity decreases the rate of second offense of breast cancer from 20 to 50 % at the women beforehand treated for breast cancer.

The objectives:

* participate as a supplement to the physiotherapist in the mobilization of the operated shoulder
* act in association with the surgical and medical team to release the adhesions superficial
* welcome these women hurt through a participative sports project
* get them a fencing adapted in a friendly atmosphere
* offer them personalized exchanges
* to propose a consequent energy expenditure but according to each and to the context
* have a practice of the operated side
* make them practise a sport with pleasure and without fatal effects

By the practice of the sports activity, investigators wish to help these people upset in their life to find the joy of life, to have projects, to find some pleasure to share moments of user-friendliness. Having led a fight against the disease to help them to lead a new fight of fencer happy to have a practice.

ELIGIBILITY:
Inclusion Criteria:

* patients operated for the breast cancer in the Hospital Rene Dubos
* patients who have sign a consent
* patients having supplied an aptitude certificate in fencing

Exclusion Criteria:

* patients who have a contraindication in the sport

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients opered for breast cancer followed at the Hospital Rene Dubos
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
quality of life questionnary | 20 sporting session, an average of one year

CONTACTS AND LOCATIONS:
Overall Officials: VAUTIER-RIT Sophie, PH, Principal Investigator — Rene Dubos Hospital

IPD SHARING:
Plan to Share IPD: No